CLINICAL TRIAL: NCT02143453
Title: Comparative Study of High Intensity Interval Training and Endurance Training in Juvenile Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Bruno Gualano, Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: HIIT in Juvenile Obesity
Record Dates: First submitted 2014-05-18; First posted 2014-05-21 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: Obesity
Keywords: exercise; overweight; children
MeSH Terms: conditions — Obesity; Motor Activity; Overweight | interventions — Endurance Training; High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High intensity interval training (Experimental)
  Interventions: Other: High intensity interval training
- Endurance training (Experimental)
  Interventions: Other: Endurance training

INTERVENTIONS:
Other: Endurance training — 30 to 60-minute continuous exercise at 80% of the peak heart rate
  Arms: Endurance training
Other: High intensity interval training — 3 to 6 sets of 60-second sprints at 100% of the peak velocity interspersed by a 3-min active recovery period.
  Arms: High intensity interval training

SUMMARY:
Exercise is an effective strategy to manage juvenile obesity; however this ideal exercise training mode is still unclear. In this study, the investigators compared the health-related effects of high intensity interval training versus endurance training in obese children.

ELIGIBILITY:
Inclusion Criteria:

* age between 8 and 12 years
* Body mass index (BMI) = 95th percentile, according to the First National Health and Nutrition Examination Survey
* no pharmacological treatment
* no evidence of metabolic, hormonal, orthopedic, and cardiovascular disease at the time of the study's commencement
* no participation in any regular exercise training program (except physical education classes, two days a week) at least 6 months before the commencement of the study and throughout the protocol.

Exclusion Criteria:

* non-obese participants
* physically active participants
* participants with cardiovascular diseases or any other condition that could preclude the participation in the the exercise training program

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2010-08; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
body mass index (BMI) | 12 weeks
aerobic conditioning (VO2max) | 12 weeks
insulin sensitivity (HOMA-index) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Gualano, Professor, Principal Investigator — University of Sao Paulo
Locations (1):
- General Hospital (School of Medicine, University of Sao Paulo), São Paulo, São Paulo, Brazil